CLINICAL TRIAL: NCT04259320
Title: Effect of the Use of Beeswax-containing Barrier on the Prevention of Nipple Crack in Lactating Primiparous Women Within the First 24 Hours After Giving the Birth: A Randomized Controlled Trial
Brief Title: The Effect of the Beeswax-containing Barrier on the Prevention of Nipple Crack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Karabuk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seda Serhatlioglu, Principal Investigator, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-01
Record Dates: First submitted 2020-02-02; First posted 2020-02-06 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Breastfeeding; Cracked Nipple in Puerperium
MeSH Terms: conditions — Breast Feeding | interventions — Milk, Human

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beeswax containing barrier (Experimental): Beeswax containing barrier will be given to the breastfeeding mother within the first 24 hours. After breastfeeding, it can be placed on the breast after it is expected to dry a little.Outside of breastfeeding and bathing, it will be constantly attached to the breasts.
  Interventions: Device: Beeswax containing barrier
- Breast milk (Experimental): After breastfeeding, 2-3 drops of breast milk are applied to the nipple and areola. After the milk has dried, the breasts are closed. This application should be done at least 5 times a day.
  Interventions: Biological: Breast milk
- No treatment- control (No Intervention): It is a group that does not use any method to prevent nipple cracks. All follow-ups in the experimental groups are done.

INTERVENTIONS:
Device: Beeswax containing barrier — Use beeswax containing barrier on each nipple after each breastfeeding.
  Arms: Beeswax containing barrier
Biological: Breast milk — Apply breast milk on each nipple and areola after each breastfeeding.
  Arms: Breast milk

SUMMARY:
In the planned study, it was aimed to evaluate the effectiveness of the beeswax-containing barrier and breast milk used in the first ten days of breastfeeding to prevent the formation of nipple cracks. It's a prospective, randomized study based on 90 primipara lactating women. Participants were assigned randomly 3 groups (beeswax-containing barrier, breast milk, and no treatment-control).

DETAILED DESCRIPTION:
Current evidence-based guidelines report that the incidence of nipple cracks ranges between 34-96%. Nipple cracks generally occur in the first week after the birth and may continue in the following periods of breastfeeding. Nipple crack is the second most common reason to stop breastfeeding early, after perceived insufficient milk release. Nipple crack pain in studies has been expressed as extremely painful and terrible. It is known that breast milk, olive oil, quince seed jelly, mint juice, lanolin, jujube fruit lotion, guaiazulen pomade, aloe vera gel, menthol essence, vitamin A-E, curcumin extract, hydrogel dressings are recommended to mothers to prevent nipple cracks during breastfeeding. The prevention of nipple cracks, will successfully allow to continue breastfeeding. In this way, breastfeeding will not be interrupted and the rate of breastfeeding-only feeding will increase in the first 6 months. Using non-pharmacological, effective and therapeutic methods will also have a positive effect to increase the rate of breastfeeding.

Studies in the literature cover the evaluation of the effectiveness of beeswax or beeswax-containing mixtures on wound, burn and crack healing. Due to its natural composition with antioxidant, antimicrobial, and antiulcerative properties, beeswax is thought to be an effective and sufficient material in preventing and healing nipple cracks.

In this study, it is planned to include 90 lactating women (30 women in each group) to meet the parametric test assumptions in the experimental and control groups (beeswax-containing barrier, breast milk, and no treatment-control). Breastfeeding mothers to be included in the experimental and control groups will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old;
* Normal spontaneous delivery.
* Pregnancy weeks between 37-42.
* Single birth.
* Initiated breastfeeding.
* Having given birth to a healthy, full-term child.
* Newborn with no oral, palatal or maxillofacial abnormalities.
* Not taking any medication, considering that drug use may cause nipple problems.
* Being able to read and write.
* Volunteering to participate in the study.
* Not having contraindications for breastfeeding.

Exclusion Criteria:

* Not approving to participate in the research.
* Being a multipara.
* Not breastfeeding within the first 24 hours.
* Development of any breast problem: Mastitis, engorgement etc.
* Taking newborn into intensive care.
* Not sticking to the application.
* Using another nipple crack preventing method during application.
* Being allergic to beeswax.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — primipara lactating women who is in the first ten days of breastfeeding
Enrollment: 90 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Nipple crack change | Change from baseline nipple crack at 10 days
  Use Nipple Crack score 0-3 (Nipple cracks increase as the score increases)

SECONDARY OUTCOMES:
Severity of nipple pain change | Change from baseline severity of nipple pain at 10 days.
  Use Numeric Rating Scale 0-10 point (The severity of pain increases as the score increases)

OTHER OUTCOMES:
Presence of nipple pain change | Change from baseline presence of nipple pain at 10 days.
  Questionary (Yes/No)
Maternal satisfaction | Baseline from baseline nipple crack at 10 days
  Questionary (Use the satisfaction categories-likert)

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Mutlu, OB/GYN, Study Director — Karabuk University Research and Training Hospital
Locations (1):
- Karabuk University Training and Research Hospital, Karabük, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After begin to study

REFERENCES:
- [Background] Buck ML, Amir LH, Cullinane M, Donath SM; CASTLE Study Team. Nipple pain, damage, and vasospasm in the first 8 weeks postpartum. Breastfeed Med. 2014 Mar;9(2):56-62. doi: 10.1089/bfm.2013.0106. Epub 2013 Dec 31. PMID 24380583
- [Background] Puapornpong P, Paritakul P, Suksamarnwong M, Srisuwan S, Ketsuwan S. Nipple Pain Incidence, the Predisposing Factors, the Recovery Period After Care Management, and the Exclusive Breastfeeding Outcome. Breastfeed Med. 2017 Apr;12:169-173. doi: 10.1089/bfm.2016.0194. Epub 2017 Mar 9. PMID 28278382
- [Background] Dennis CL, Jackson K, Watson J. Interventions for treating painful nipples among breastfeeding women. Cochrane Database Syst Rev. 2014 Dec 15;2014(12):CD007366. doi: 10.1002/14651858.CD007366.pub2. PMID 25506813
- [Derived] Serhatlioglu S, Gencturk N, Mutlu S. Determination of the effectiveness of beeswax in preventing nipple pain and cracks in primiparous breastfeeding mothers: A randomized controlled trial. Explore (NY). 2023 Nov-Dec;19(6):851-858. doi: 10.1016/j.explore.2023.05.002. Epub 2023 May 13. PMID 37236877